CLINICAL TRIAL: NCT03035552
Title: Randomized Controlled Trial to Improve Oral Feeding Outcomes in Infants With Complex Congenital Heart Disease Using Pacifier Activated Device-Training With Mother's Voice
Brief Title: CTICU Pacifier Activated Music Player and Mother's Voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Kristen Benninger, MD, MD, PhD, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB16-00493
Record Dates: First submitted 2017-01-23; First posted 2017-01-30 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Heart Defects, Congenital
Keywords: Congenital heart disease (CCHD); Non-Nutritive Suck
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Randomized to Pacifier Activated Lullaby (mother's voice contingent on suck, 15 minutes, 5 sessions) before surgery or and Sounds of Love (mother's voice playing freely, 15 minutes, 5 sessions). Arm 2: Sounds of love before surgery, Pacifier activated lullaby after the surgery.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessors and the investigator are masked to the group assignment
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment prior to surgery (Experimental): Infants randomized to receive the pacifier activated music player and mother's voice treatment prior to surgery for 5 sessions, and mother's voice playing freely post surgery.
  Interventions: Behavioral: Pacifier activated music player
- Treatment post surgery (Experimental): Infants randomized to receive the mother's voice playing freely prior to surgery,and pacifier activated music player and mother's voice treatment post surgery for 5 sessions.
  Interventions: Behavioral: Pacifier activated music player

INTERVENTIONS:
Behavioral: Pacifier activated music player — Therefore the immediate goal of the current proposal is to demonstrate that intensive NNS-training using reinforcement with mother's voice can improve the oral feeding outcomes of infants with CCHD using a randomized controlled trial (RCT) design, with wait-list controls to ensure that infants in the trial all benefit from a treatment with only demonstrated positive effects. Establishment of optimal NNS patterns in the first 6 months after birth in these infants will improve downstream feeding skills and may promote better motor and language outcomes by one year of age.
  Other Names: PAM

SUMMARY:
The purpose of this study is to determine if intensive training of Non-Nutritive Suck (NNS) using contingent positive reinforcement with mother's voice can improve the feeding outcomes of infants with congenital heart defect (CHD) at high risk for oral motor problems.

DETAILED DESCRIPTION:
Randomized controlled trial to Improve Oral Feeding Outcomes in Infants with Complex Congenital heart disease using Pacifier Activated Device-Training with Mother's Voice Specific Aims Infants with complex congenital heart disease (CCHD) have high rates of delayed or impaired oral feeding skills, associated with other neurodevelopmental problems such as worse motor and language outcomes in early childhood. The acquisition of efficient suck strength and patterns is essential to promote later optimal oral feeding. Therefore, ineffective non-nutritive suck (NNS), one of the earliest feeding milestones, can result in later maladaptive oral motor skills or even oro-sensory aversions. Evidence-based interventions are lacking for CCHD infants hospitalized in the Cardiothoracic Intensive Care Unit (CTICU) to improve early oral feeding patterns and promote acquisition of later developmental milestones. NNS training (as opposed to simply offering a pacifier) safely improves oral feeding strength and rate in other high-risk populations, such as preterm infants, even when they have suffered severe neural insults. This type of training uses operant conditioning with positive stimuli to reinforce learning and establishment of functional pathways between lower and higher order neural networks. Furthermore, NNS training is associated with acquisition of essential developmental milestones in the first year. The investigators propose the following hypothesis: Intensive NNS-contingent training using reinforcement with mother's voice can improve the oral feeding outcomes of infants with CCHD. They further hypothesize that establishment of optimal NNS in the first 6 months can improve feeding and developmental outcomes by one year of age.

To test this hypothesis, the investigators propose a randomized controlled trial (RCT) in CCHD infants hospitalized for surgical repair. Because the proposed intervention has been demonstrated to only have positive effects in other high-risk infants, the study will use a wait-list design: CCHD infants who do not receive their intervention before surgery will receive it after, so that the entire cohort will eventually benefit from the intervention. The intervention will utilize a Pacifier Activated Music Player (PAM) with a sensor detecting changes in suck pressures and patterns, and a speaker contingently delivering mother's voice, in infants 0-6 months in the CTICU. Quantitative oral feeding metrics before and after the intervention, as well as, immediately after discharge will be used to measure efficacy. Secondly, to assess the impact of NNS training on developmental milestone acquisition, a standardized feeding and neurodevelopmental assessments of all trial infants at 12 months of age in the Follow-Up clinic will also be conducted. Randomization will account for differences in CCHD diagnoses known to impact outcomes. The study design will control for the type of surgical procedure as a proxy for severity of illness and exposure to anesthesia and for variables associated with neurodevelopment such as maternal education and prematurity.

Aim 1 A: Compare oral feeding skills as measured by suck strength, rate and burst patterns in CCHD infants with vs. without NNS training using PAM/mother's voice prior to surgery, in an RCT design. Aim 1 B: Correlate improvements in oral feeding skills after NNS training with PAM/mother's voice in the entire study cohort with higher scores on standardized feeding questionnaires at 1 month after discharge. Aim 2: Demonstrate that improvements in oral feeding skills in the CTICU will correlate with better neurodevelopmental outcomes as measured by standardized scores on the Bayley Scales of Infant and Toddler Development (BSID III) at 12 months. This study holds significant public health relevance as it validates an inexpensive, parent-centered rehabilitative strategy for infants at high-risk for impaired oral feeding skills, with a device and approach easily adapted to many levels of CCHD care and with the potential to improve longer-term neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* Infants that have a diagnosis of a complex congenital heart defect and scheduled for a surgical intervention; meet CTICU feeding guidelines criteria. Infants with acquired brain injury will be included, as well as those whose mothers speak languages other than English.

Exclusion Criteria:

* Infants that are on assisted ventilation, continuous positive airway pressure, general anesthesia within 24 hours; lethal congenital abnormalities or congenital brain malformation.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Oral feeding Efficiency | Depending on randomization, 5 days pre-operation (group 1) or 5 days post-operation (group 2)
  Continuous measure of suck strength and suck rate during oral feeding via PAM sensor, as well as suck burst pattern and average oral feeding volumes.

SECONDARY OUTCOMES:
Oral feeding development | Thirty days post-operation
  Analyzing individual milestones via the American Speech-Language-Hearing Association assessment by speech language pathology, and adverse feeding events.
Neurodevelopment | Twelve months
  Evaluating participant's development using Bayley Scales of Infant and Toddler Development (BSID III)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Maitre, MD. PhD, Principal Investigator — Perinatal Research Institute, Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411
- [Background] Brosig C, Mussatto K, Hoffman G, Hoffmann RG, Dasgupta M, Tweddell J, Ghanayem N. Neurodevelopmental outcomes for children with hypoplastic left heart syndrome at the age of 5 years. Pediatr Cardiol. 2013 Oct;34(7):1597-604. doi: 10.1007/s00246-013-0679-3. Epub 2013 Mar 16. PMID 23503929
- [Background] Walker K, Badawi N, Halliday R, Stewart J, Sholler GF, Winlaw DS, Sherwood M, Holland AJ. Early developmental outcomes following major noncardiac and cardiac surgery in term infants: a population-based study. J Pediatr. 2012 Oct;161(4):748-752.e1. doi: 10.1016/j.jpeds.2012.03.044. Epub 2012 May 10. PMID 22578999
- [Background] Luyckx K, Missotten L, Goossens E, Moons P; i-DETACH Investigators. Individual and contextual determinants of quality of life in adolescents with congenital heart disease. J Adolesc Health. 2012 Aug;51(2):122-8. doi: 10.1016/j.jadohealth.2011.11.007. Epub 2012 Feb 22. PMID 22824441
- [Background] Cassidy AR, White MT, DeMaso DR, Newburger JW, Bellinger DC. Executive Function in Children and Adolescents with Critical Cyanotic Congenital Heart Disease. J Int Neuropsychol Soc. 2015 Jan;21(1):34-49. doi: 10.1017/S1355617714001027. Epub 2014 Dec 9. PMID 25487044
- [Background] Jackson JL, Misiti B, Bridge JA, Daniels CJ, Vannatta K. Emotional functioning of adolescents and adults with congenital heart disease: a meta-analysis. Congenit Heart Dis. 2015 Jan-Feb;10(1):2-12. doi: 10.1111/chd.12178. Epub 2014 Feb 26. PMID 24612910
- [Background] Adams-Chapman I, Bann CM, Vaucher YE, Stoll BJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Association between feeding difficulties and language delay in preterm infants using Bayley Scales of Infant Development-Third Edition. J Pediatr. 2013 Sep;163(3):680-5.e1-3. doi: 10.1016/j.jpeds.2013.03.006. Epub 2013 Apr 10. PMID 23582139
- [Background] Averin K, Uzark K, Beekman RH 3rd, Willging JP, Pratt J, Manning PB. Postoperative assessment of laryngopharyngeal dysfunction in neonates after Norwood operation. Ann Thorac Surg. 2012 Oct;94(4):1257-61. doi: 10.1016/j.athoracsur.2012.01.009. Epub 2012 Mar 14. PMID 22421593
- [Background] Dewan K, Cephus C, Owczarzak V, Ocampo E. Incidence and implication of vocal fold paresis following neonatal cardiac surgery. Laryngoscope. 2012 Dec;122(12):2781-5. doi: 10.1002/lary.23575. Epub 2012 Sep 5. PMID 22952115
- [Background] Sachdeva R, Hussain E, Moss MM, Schmitz ML, Ray RM, Imamura M, Jaquiss RD. Vocal cord dysfunction and feeding difficulties after pediatric cardiovascular surgery. J Pediatr. 2007 Sep;151(3):312-5, 315.e1-2. doi: 10.1016/j.jpeds.2007.03.014. Epub 2007 Jun 26. PMID 17719946
- [Background] Davies RR, Carver SW, Schmidt R, Keskeny H, Hoch J, Pizarro C. Laryngopharyngeal dysfunction independent of vocal fold palsy in infants after aortic arch interventions. J Thorac Cardiovasc Surg. 2014 Aug;148(2):617-24.e2. doi: 10.1016/j.jtcvs.2013.05.054. Epub 2013 Nov 26. PMID 24290573
- [Background] Limperopoulos C, Majnemer A, Shevell MI, Rosenblatt B, Rohlicek C, Tchervenkov C. Neurodevelopmental status of newborns and infants with congenital heart defects before and after open heart surgery. J Pediatr. 2000 Nov;137(5):638-45. doi: 10.1067/mpd.2000.109152. PMID 11060529
- [Background] Pereira Kda R, Firpo C, Gasparin M, Teixeira AR, Dornelles S, Bacaltchuk T, Levy DS. Evaluation of swallowing in infants with congenital heart defect. Int Arch Otorhinolaryngol. 2015 Jan;19(1):55-60. doi: 10.1055/s-0034-1384687. Epub 2014 Nov 5. PMID 25992152
- [Background] Skinner ML, Halstead LA, Rubinstein CS, Atz AM, Andrews D, Bradley SM. Laryngopharyngeal dysfunction after the Norwood procedure. J Thorac Cardiovasc Surg. 2005 Nov;130(5):1293-301. doi: 10.1016/j.jtcvs.2005.07.013. Epub 2005 Oct 13. PMID 16256781
- [Derived] Kjeldsen CP, Emery L, Simsic J, He Z, Stark AR, Neel ML, Maitre NL. Contingent Mother's Voice Intervention Targeting Feeding in Hospitalized Infants with Critical Congenital Heart Defects. Children (Basel). 2023 Sep 30;10(10):1642. doi: 10.3390/children10101642. PMID 37892305